CLINICAL TRIAL: NCT03098628
Title: Trial of Simplified Pneumococcal Vaccination in Vietnam II: The Herd Immunity Approach
Brief Title: Trial of Simplified Pneumococcal Vaccination in Vietnam II
Acronym: VPTII
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Pasteur Institute, Ho Chi Minh City (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HREC36027
Record Dates: First submitted 2017-03-01; First posted 2017-04-04 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2023-08

CONDITIONS: Pneumococcal Vaccine
MeSH Terms: interventions — five-valent pneumococcal conjugate vaccine

STUDY DESIGN:
Intervention Model Description: single-blind, open-label, randomised controlled trial
Who Masked: Outcomes Assessor
Masking Description: This is a single-blind, open-label, randomised trial, with laboratory staff blinded to study group allocation as all the outcome measures that address the study objectives are laboratory based. Laboratory samples will be labelled with a unique trial identification number that does not identify the study group. Given the different timing of the vaccine schedules in the different study arms, the study nurses, vaccine administrators and participants will not be blinded to the study group allocation of each infant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- V - PCV10 vaccine, 0+1 (Active Comparator): PCV10, 0+1 schedule. PCV vaccine at 12 months of age
  Interventions: Biological: PCV Vaccine
- W - PCV13 vaccine, 0+1 (Active Comparator): PCV13 in 0+1 schedule. PCV vaccine at 12 months of age
  Interventions: Biological: PCV Vaccine
- X - PCV10 vaccine, 1+1 (Active Comparator): PCV10, 1+1 schedule. PCV vaccine given at 2 and 12 months of age
  Interventions: Biological: PCV Vaccine
- Y - PCV13 vaccine, 1+1 (Active Comparator): PCV13, 1+1 schedule. PCV vaccine at 2 and 12 months of age
  Interventions: Biological: PCV Vaccine
- Z - Control (Other): Control group. PCV vaccine given at end of study (24 months)
  Interventions: Biological: PCV Vaccine

INTERVENTIONS:
Biological: PCV Vaccine — PCV vaccination

SUMMARY:
This is a single-blind, open-label, randomised controlled trial with five groups. There are four different Pneumococcal Conjugate Vaccine (PCV) schedules to be evaluated.

DETAILED DESCRIPTION:
This is a single-blind, open-label, randomised controlled trial with five groups. There are four different PCV schedules to be evaluated: a 0+1 schedule of PCV10 at 12 months of age (Group V), a 0+1 schedule of PCV13 at 12 months of age (Group W), a 1+1 schedule of PCV10 at 2 and 12 months of age (Group X), and a 1+1 schedule of PCV13 at 2 and 12 months of age (Group Y); along with a control group that receives a dose of PCV10 at 24 months of age (Group Z). Additionally, all participants will receive four doses of Infanrix-hexa at 2, 3, 4 and 18 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 2 months and 2 months plus 2 weeks;
* No significant maternal or perinatal history;
* Born at or after 36 weeks gestation;
* Written and signed informed consent from parent/legal guardian;
* Lives within approximately 30 minutes of the commune health centre;
* Family anticipates living in the study area for the next 22 months

Exclusion Criteria:

* Known allergy to any component of the vaccine;
* Allergic reaction or anaphylactic reaction to any previous vaccine;
* Known immunodeficiency disorder;
* Known HIV-infected mother;
* Known thrombocytopenia or coagulation disorder;
* Administration or planned administration of any immunoglobulin or blood product since birth;
* Severe birth defect requiring ongoing medical care;
* Chronic or progressive disease;
* Seizure disorder;
* History of severe illness;
* Receipt of any 2 month vaccines through the Expanded Programme of Immunization (EPI) program;
* Family plans on giving the infant Quinvaxem (DTP-Hib-HBV).

Additionally, enrolment will be deferred and infants asked to return to the health centre one week later for reassessment if they have at least one of the following deferral criteria:

* Axillary temperature ≥37.5°C or ≤35.5°C;
* Acute infection, especially bacterial;
* Oral administration of corticoid therapy in past 14 days; or
* Any of the following symptoms that interfere with normal activities: crying more than usual, sleeping more than usual, or loss of appetite.

Ages: 8 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2501 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-06-11 (Actual)

PRIMARY OUTCOMES:
Carriage of Vaccine Type pneumococci | 12 months post vaccination, i.e. 24 months of age
  Evaluate the effect of a 0+1 PCV schedule administered at 12 months of age on Nasopharngeal Carrige (NP) carriage during the first two years of life, comparing a) PCV10-vaccinated and b) PCV13-vaccinated participants with unvaccinated controls
Carriage of Vaccine Type pneumococci | 12 months post last vaccination, i.e. 24 months of age
  Evaluate the effect of a 1+1 PCV schedule administered at 2 and 12 months of age on NP carriage during the first two years of life, comparing a) PCV10-vaccinated and b) PCV13-vaccinated participants with unvaccinated controls.

SECONDARY OUTCOMES:
Immunology sub-study | 12 months post vaccination, i.e. 24 months of age
  i) To evaluate the immune responses to a 0+1 PCV schedule at 12 months of age, comparing a) PCV10-vaccinated and b) PCV13-vaccinated participants with unvaccinated controls;
Immunology sub-study | 12 months post last vaccination, i.e. 24 months of age
  ii) To evaluate the immune responses to a 1+1 PCV schedule at 2 and 12 months of age, comparing a) PCV10-vaccinated and b) PCV13-vaccinated participants with unvaccinated controls;

CONTACTS AND LOCATIONS:
Overall Officials: Kim Mulholland, MD, Principal Investigator — Murdoch Childrens Research Institute; Nguyen Vu Thuong, MD, Principal Investigator — Pasteur Institute
Locations (1):
- Pasteur Institute, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Temple B, Tran HP, Dai VTT, Smith-Vaughan H; VPT-II Collaborator Group; Licciardi PV, Satzke C, Nguyen TV, Mulholland K. Efficacy against pneumococcal carriage and the immunogenicity of reduced-dose (0 + 1 and 1 + 1) PCV10 and PCV13 schedules in Ho Chi Minh City, Viet Nam: a parallel, single-blind, randomised controlled trial. Lancet Infect Dis. 2023 Aug;23(8):933-944. doi: 10.1016/S1473-3099(23)00061-0. Epub 2023 Apr 14. PMID 37062304
- [Derived] Temple B, Tran HP, Dai VTT, Bright K, Uyen DY, Balloch A, Licciardi P, Nguyen CD, Satzke C, Smith-Vaughan H, Nguyen TV, Mulholland K. Simplified 0+1 and 1+1 pneumococcal vaccine schedules in Ho Chi Minh City, Vietnam: protocol for a randomised controlled trial. BMJ Open. 2021 Nov 29;11(11):e056505. doi: 10.1136/bmjopen-2021-056505. PMID 34845082